CLINICAL TRIAL: NCT04037761
Title: Shanghai Children's Health, Education and Lifestyle Evaluation, Preschool (the SCHEDULE-P) Cohort Study
Brief Title: Shanghai Children's Health, Education and Lifestyle Evaluation, Preschool (the SCHEDULE-P Study)
Status: Recruiting | Type: Observational
Sponsor: Sijia Gu (Other)
Responsible Party: Sponsor-Investigator, Sijia Gu, Responsible Party, Clinical Research, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: SCMCIRB-K2016022-01
Record Dates: First submitted 2019-06-25; First posted 2019-07-30 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Child Development
Keywords: early child development; cohort study; education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shanghai is one of pilot areas for the early education of 3-6 years old infants in China. Shanghai Municipal Education Commission has been actively exploring more effective early education guidance methods. This survey, in the form of online questionnaire and site test, aims to dynamically evaluate the changes in the early development level of children in Shanghai and provide scientific basis for providing better early education services in the future.

ELIGIBILITY:
Inclusion Criteria:

* All 3-year-old children entered into public kindergartens or private kindergartens in Shanghai since 2016.

Exclusion Criteria:

* Children entered into international kindergartens

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A stratified random sample of children aged 3-4 from 9 levels kindergartens in 16 districts of Shanghai.
Sampling Method: Probability Sample
Enrollment: 20899 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Demographics and Socioeconomic statue information | 2 weeks
  Including parent's education, family income, etc.
Child Care Environment | 2 weeks
  The ICCE measures child care environment through 13 questions in four subscales: "human stimulation" , "social stimulation", "avoidance of restriction", and "social support". It can be used as a self-report or interview, meaning that it does not necessarily need a home visit. Each item is assessed using a multiple-choice format, and the answer is given a binary score according to the manual (1 = good, 0 = not good or not sure); the overall score is calculated by summing all items in the scale. A higher score indicates a better child care environment.
Parent-child interaction | 2 weeks
  Chinese parent-child interaction scale (CPCIS): Parent-child interaction was assessed using the Chinese Parent-Child Interaction Scale, a standardized questionnaire, which has been well-validated using Rasch analysis. It has also been shown to have good person-separation reliability (0.82). Parents were asked to indicate the frequency of 12 parent-child interactive activities they engaged in during the past month on a scale of 0-5 (0 = not occurring, 5 = very frequent). The questionnaire measures the quantity of the most common activities of learning related, reading, recreation, and interaction with environment. The total scores added from all activities were used in the analysis.
Child behavior assessment, Sleep Habits | 2 weeks
  Children's Sleep Habits Questionnaire (CHSQ) Sleep onset and wake up time in the past weekdays and weekends were collected from a parent reported Children Sleep Habits Questionnaire23 and sleep duration in weekdays and weekends was calculated separately. Daily average sleep duration was calculated using the formula: ([weekday sleep duration×5] + [weekend sleep duration×2])/7.
Child behavior assessment, Screening Exposure | 2 weeks
  Parents according to the situation of children over the past month, respectively report children's school day and rest every day to watch quiz and educational video programs, entertainment, the children watch every day and educational video programs, entertainment, the children every day to watch video programs, entertainment, the children's television, playing video games, and playing video games and browsing the web time.
Early Child Development | 2 weeks
  We perform Early Human Capability Index (eHCI) to evaluate early childhood development in 3-5-year-olds that predicts future capabilities. It covers general verbal communication, approaches to learning, numeracy and concepts, formal literacy-reading and writing, cultural knowledge, social and emotional skills, perseverance, and physical health of child development. For each domain, the scores range from 0 through to 1, with 1 being the best score and 0 the worst.
Social-emotion | 2 weeks
  The Strengths and Difficulties Questionnaire (SDQ) we use in this survey is a short screening questionnaire covering the current difficulties in social psychology (i.e. emotional symptoms, conduct problems, hyperactivity-inattention, peer problems), and personal strengths (i.e. prosocial behavior). High SDQ score is associated with an increase in psychiatric risk, on the opposite, prosocial behavior score is positive with prosocial behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China